CLINICAL TRIAL: NCT02985151
Title: A Single Center, Double-blinded Randomized Placebo-controlled Trial to Evaluate Surgical Scars After Treatment With Fractional Carbon Dioxide Rejuvenation Laser Therapy
Brief Title: Interventional Study to Evaluate the Appearance of Surgical Scars After Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Ramona Behshad, MD, Associate Professor, Department of Dermatology, St. Louis University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SLU-27403
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Cicatrix; Carbon Dioxide Laser
Keywords: Scar; Carbon Dioxide Laser; Laser Ablation
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: This is a crossover study where subjects are randomized into two arms. Subjects in the sham arm are allowed to crossover at the end of their initial intervention period.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- High Energy Treatment Group (Active Comparator): Subjects in this group will receive at least two Syneron-Candela CO2RE laser treatments set at either the Mid mode or the Deep mode of the laser at visits three months apart. Thereafter, individuals in this group will be offered a third optional treatment at one of these settings.
  Interventions: Device: Syneron-Candela CO2RE Laser
- Low Energy Placebo Group (Placebo Comparator): Subjects in this group will receive at least two Syneron-Candela CO2RE laser treatments set at the Light mode of the laser at visits three months apart. The Light mode is a low energy setting that superficially cleanses the skin, and would not affect the scar, which is deeper in the skin. Individuals in this group will be offered two optional high energy treatments subsequent to receiving the two light energy treatments.
  Interventions: Device: Syneron-Candela CO2RE Laser

INTERVENTIONS:
Device: Syneron-Candela CO2RE Laser — This fractionated ablative laser will administer energy at either a high intensity setting or a low intensity setting to subjects randomized into a particular treatment group. It will be operated by the principle investigator, who has extensive experience with laser therapy.

SUMMARY:
This study evaluates the effect of a fractionated carbon dioxide laser on surgical scars of the face and neck over 12 months. Anyone with a surgical scar on the face and neck who has not had laser therapy may be eligible to participate. The visits occur every three months for up to 12 months. Subjects will be randomly assigned to receive a higher energy treatment or a lower energy treatment during the study. Subjects and raters will be blinded to which therapy level the patient receives. At each visit, the scars will be photographed and the subject will complete a questionnaire to rate the scar prior to treatment. Three physicians will evaluate the scar at each visit. One rater will evaluate the scars in person during the visit, while the other two raters will evaluate the scars using photographs after each visit. During the first three study visits, subjects will receive their assigned treatment, obtain post-treatment instructions, and a diary to record redness, swelling, pain, itching, or other skin changes after treatment. At the third study visit, subjects will have the option to receive additional treatments or terminate their participation in the study. The fourth visit for those who continue will be a treatment visit for one group and the fifth visit will be for data collection, with no treatment offered.

DETAILED DESCRIPTION:
In dermatology, the use of Light Amplification by Stimulated Emission of Radiation (laser) has revolutionized the management of various conditions including angiomas, vitiligo, wrinkles, and scars. (Omi, 2014 and Chapas, 2008) Scars result from sub-optimal collagen production during wound healing leading to topographical irregularities. To effectively modify these defects, any treatment must be capable of penetrating the epidermis and eliciting dermal remodeling at a depth of at least 1 mm. The 10,600 nm carbon dioxide (CO2) laser utilizes high energy at short durations to vaporize intra- and extra-cellular water, resulting in tissue ablation causing a substantial thermal injury to the dermis, reducing the likelihood of additional scarring. The CO2 laser can stimulate collagen production and theoretically improve scar thickness, pliability, and texture.

This study is a prospective, randomized double-blinded placebo-controlled trial to evaluate the efficacy of fractionated carbon dioxide laser in improving surgical scars on the head and neck over 3-5 study visits for a duration of 12.5 months. Scar assessments will be based on objective changes identified on pictures taken with the Canfield Vectra M3 3D Imaging System and subjective changes identified with the Patient and Observer Scar Assessment Scale (POSAS), a validated scar scale. As a secondary objective, the study will evaluate the tolerability of the laser, by assessing the severity and duration of known side effects of laser therapy such as erythema, edema, burning sensation, post-inflammatory pigment changes, infection, scarring, xerosis, pruritus, bronzing, and any other adverse events that arise following treatment. Subjects will be given a diary after each treatment to document this information.

ELIGIBILITY:
Inclusion Criteria:

* Surgical scar present in the head or neck region for at least 8 weeks.
* Capable of providing informed consent
* Available for study appointments
* Follows directions of post-treatment instructions

Exclusion Criteria:

* Individuals under the age of 18
* Prior laser treatment to the head or neck
* History of keloid formation
* Isotretinoin use in the last 6 months prior to study enrollment
* Allergy to topical lidocaine
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramona Behshad, MD, Principal Investigator — Saint Louis University, Department of Dermatology
Locations (1):
- Saint Louis University Department of Dermatology-Des Peres Med Arts Pavilion II, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be accessed after publication of the results in a medical journal.

REFERENCES:
- [Background] Omi T, Numano K. The Role of the CO2 Laser and Fractional CO2 Laser in Dermatology. Laser Ther. 2014 Mar 27;23(1):49-60. doi: 10.5978/islsm.14-RE-01. PMID 24771971
- [Background] Bodendorf MO, Grunewald S, Wetzig T, Simon JC, Paasch U. Fractional laser skin therapy. J Dtsch Dermatol Ges. 2009 Apr;7(4):301-8. doi: 10.1111/j.1610-0387.2008.06845.x. Epub 2008 Aug 28. English, German. PMID 18761608
- [Background] Chapas AM, Brightman L, Sukal S, Hale E, Daniel D, Bernstein LJ, Geronemus RG. Successful treatment of acneiform scarring with CO2 ablative fractional resurfacing. Lasers Surg Med. 2008 Aug;40(6):381-6. doi: 10.1002/lsm.20659. PMID 18649382
- [Background] Majid I, Imran S. Fractional CO2 Laser Resurfacing as Monotherapy in the Treatment of Atrophic Facial Acne Scars. J Cutan Aesthet Surg. 2014 Apr;7(2):87-92. doi: 10.4103/0974-2077.138326. PMID 25136208
- [Background] van der Wal MB, Tuinebreijer WE, Bloemen MC, Verhaegen PD, Middelkoop E, van Zuijlen PP. Rasch analysis of the Patient and Observer Scar Assessment Scale (POSAS) in burn scars. Qual Life Res. 2012 Feb;21(1):13-23. doi: 10.1007/s11136-011-9924-5. Epub 2011 May 20. PMID 21598065
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 patients enrolled in the study. One subject withdrew from the study prior to treatment. A total of 50 subjects received treatment in the study. There were 10 subjects who crossed-over from low-energy treatment to high-energy treatment after completing the low-energy portion of the study.
Groups:
- High Energy Treatment Group: Subjects in this group received one to two Syneron-Candela CO2RE laser treatments set at either the Mid mode or the Deep mode of the laser at visits three months apart. Thereafter, individuals in this group were offered a third optional treatment at one of these settings.
  Syneron-Candela CO2RE Laser: This fractionated ablative laser will administer energy at either a high-intensity setting or a low-intensity setting to subjects randomized into a particular treatment group. It will be operated by the principal investigator, who has extensive experience with laser therapy.
- Low Energy Placebo Group: Subjects in this group were offered two optional high-energy treatments subsequent to receiving the two light-energy treatments. Syneron-Candela CO2RE laser treatments set at the Light mode of the laser at visits three months apart. The Light mode is a low-energy setting that superficially cleanses the skin, and would not affect the scar, which is deeper in the skin. Individuals in this group will be offered two optional high-energy treatments subsequent to receiving the two light-energy treatments.
  Syneron-Candela CO2RE Laser: This fractionated ablative laser administered energy at either a high-intensity setting or a low intensity setting to subjects randomized into a particular treatment group. It was operated by the principal investigator, who has extensive experience with laser therapy.
Period: Original Randomization
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Started | 25 | 26
Completed | 25 | 25
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Crossover From Low to High Energy
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Started | 0 | 10
Completed | 0 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Energy Treatment Group: Subjects in this group received one or two Syneron-Candela CO2RE laser treatments set at either the Mid mode or the Deep mode of the laser at visits three months apart. Thereafter, individuals in this group were offered a third optional treatment at one of these settings.
  Syneron-Candela CO2RE Laser: This fractionated ablative laser administered energy at either a high-intensity setting or a low intensity setting to subjects randomized into a particular treatment group. It was operated by the principal investigator, who has extensive experience with laser therapy.
- Total: Total of all reporting groups
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.7) | 56.3 (10.7) | 58.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 21 | 24 | 45
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Baseline Scar Length [Mean (Standard Deviation); unit: mm] — Visit 1 scar dimensions measured by Vectra analysis
  mm | 31.0 (17.42809) | 36.8 (27.25163) | 33.5044 (22.13543)
Baseline Scar Width [Mean (Standard Deviation); unit: mm] — Visit 1 scar dimensions measured by Vectra analysis
  mm | 10.7 (10.25) | 11.6 (9.95) | 11.08 (10.05)
Baseline Scar Surface Area [Mean (Standard Deviation); unit: cm^2] — Visit 1 scar dimensions measured by Vectra analysis
  cm^2 | 2.7 (2.37) | 4.4 (6.72) | 3.41 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Change in Vectra Measured Length V1 (Month 0)-V2 (Month 3) for Original Group; Visit 3 (Month 6) to Visit 4 (Month 9) for Crossover Group
Description: Utilizing the Vectra microtopographic imaging system, the study team will measure changes in the length of the scar after laser therapy.
Time Frame: 3 months (month 0-3 for original randomized group, month 6-9 for crossover group)
Population: The high-energy treatment group includes the 25 participants originally randomized to high-energy treatment and the 10 crossover subjects. The low-energy placebo group includes the 25 subjects who did not withdraw from the study (26 were originally randomized, and one withdrew).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
mm | 0.10 (0.78) | 0.03 (0.26)

2. Primary Outcome: In Person Blinded Observer POSAS Change V1 (Month 0)-V2 (Month 3) for Original Group; Visit 3 (Month 6) to Visit 4 (Month 9) for Crossover Group
Description: Utilizing the Patient and Observer Scar Assessment Scale (POSAS) (a scar assessment scale), the study will evaluate features of color change, thickness, width, the texture of the scar, pain associated with the scar, and itching associated with the scar by blinded clinical evaluators. Scale is scored from 1-10 with higher scores indicating a worse scar. A change in the total score is being reported.
Time Frame: 3 months (month 0-3 for original randomized group, month 6-9 for crossover group)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
score on a scale | -3.29 (3.95) | -3.30 (3.76)

3. Primary Outcome: Change in Vectra Measured Width V1 (Month 0)-V2 (Month 3) for Original Group; Visit 3 (Month 6) to Visit 4 (Month 9) for Crossover Group
Description: Utilizing the Vectra microtopographic imaging system, the study team will measure changes in the width of the scar after laser therapy.
Time Frame: 3 months (months 0-3 for the original randomized group, months 6-9 for the crossover group)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
mm | 0.06 (0.34) | -0.08 (0.39)

4. Primary Outcome: Change in Vectra Measured Surface Area V1 (Month 0)-V2 (Month 3) for the Original Group; Visit 3 (Month 6) to Visit 4 (Month 9) for Crossover Group
Description: Utilizing the Vectra microtopographic imaging system, the study team will measure changes in the surface area of the scar after laser therapy.
Time Frame: 3 months (months 0-3 for the original randomized group, months 6-9 for the crossover group)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
cm^2 | 0.01 (0.11) | -0.04 (0.15)

5. Primary Outcome: Change in Vectra Measured Length V1 (Month 0)-V3 (Month 6) for the Original Group; Visit 3 (Month 6) to Visit 5 (Month 12) for Crossover Group
Description: as for outcome 1
Time Frame: 6 months (months 0-6 for the original randomized group, months 6-12 for the crossover group)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
mm | 0.42 (1.18) | -0.23 (0.96)

6. Primary Outcome: Change in Vectra Measured Width V1 (Month 0)-V3 (Month 6) for the Original Group; Visit 3 (Month 6) to Visit 5 (Month 12) for Crossover Group
Description: as for outcome 3
Time Frame: 6 months (months 0-6 for the original randomized group, months 6-12 for the crossover group)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
mm | 0.19 (0.83) | -1.37 (4.62)

7. Primary Outcome: Change in Vectra Measured Surface Area V1 (Month 0)-V3 (Month 6) for the Original Group; Visit 3 (Month 6) to Visit 5 (Month 12) for Crossover Group
Description: Utilizing the Vectra microtopographic imaging system, the study team will measure changes in the suface area of the scar after laser therapy.
Time Frame: 6 months (months 0-6 for the original randomized group, months 6-12 for the crossover group)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
cm^2 | 0.08 (0.18) | -0.05 (0.16)

8. Primary Outcome: In-person Blinded Observer Change POSAS V1 (Month 0)-V3 (Month 6) for the Original Group; Visit 3 (Month 6) to Visit 5 (Month 12) for Crossover Group
Description: as for outcome 2
Time Frame: 6 months (months 0-6 for the original randomized group, months 6-12 for the crossover group)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
score on a scale | -4.95 (2.98) | -5.16 (5.29)

9. Primary Outcome: Change in Blinded Photo Observer Score POSAS V1 (Month 0)-V2 (Month 3) for the Original Group; Visit 3 (Month 6) to Visit 4 (Month 9) for Crossover Group
Description: Utilizing the Patient and Observer Scar Assessment Scale (POSAS) (a scar assessment scale), the study will evaluate features of color change, thickness, width, the texture of the scar, pain associated with the scar, and itching associated with the scar by the blinded clinical evaluators. Scale is scored from 1-10 with higher scores indicating a worse scar. A change in the total score is being reported.
Time Frame: 3 months (months 0-3 for the original randomized group, months 6-9 for the crossover group)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
score on a scale | -2.36 (3.51) | -2.73 (2.81)

10. Primary Outcome: Change in Blinded Photo Observer Score on POSAS V1 (Month 0)-V3 (Month 6) for the Original Group; Visit 3 (Month 6) to Visit 5 (Month 12) for Crossover Group
Description: as for outcome 2
Time Frame: 6 months (months 0-6 for the original randomized group, months 6-12 for the crossover group)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
score on a scale | -4.18 (4.38) | -4.28 (3.40)

11. Secondary Outcome: Tolerability Associated With the Laser Treatment at V1 (Month 0) and V2 (Month 3) for the Original Group; Visit 3 (Month 6) and Visit 4 (Month 9) for Crossover Group
Description: Participants will be given a diary to record the severity and duration of symptoms for the day of treatment and then daily for seven days after each laser treatment: redness, scaling/flaking, pustules, swelling, pain, itching, burning, color changes (darkening and/or lightning), infection, and any other adverse events that arise following treatment. Subjects score each of the symptom severity on a scale of 0-4 (0=none, 1= mild, 2= moderate, 3= intense, 4= intolerable). The average weekly score for each group is reported below.
Time Frame: V1 (month 0) and V2 (month 3) for the original group; visit 3 (month 6) and visit 4 (month 9) for crossover group
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
Number analyzed (Participants) | 35 | 25
score on a scale
  Patient Diary Redness After Visit 1 | 1.91 (0.73) | 1.98 (0.63)
  Patient Diary Scaling After Visit 1 | 0.58 (0.62) | 0.70 (0.53)
  Patient Diary Pustules After Visit 1 | 0.41 (0.67) | 0.29 (0.48)
  Patient Diary Swelling After Visit 1 | 1.03 (0.90) | 0.99 (0.92)
  Patient Diary Pain After Visit 1 | 0.45 (0.54) | 0.62 (0.60)
  Patient Diary Itch After Visit 1 | 0.63 (0.59) | 0.64 (0.73)
  Patient Diary Burn After Visit 1 | 0.36 (0.44) | 0.59 (0.44)
  Patient Diary Color After Visit 1 | 0.69 (0.90) | 0.95 (0.96)
  Patient Diary Infection After Visit 1 | 0.06 (0.19) | 0.0 (0.0)
  Patient Diary Redness After Visit 2 | 1.78 (0.77) | 2.00 (0.62)
  Patient Diary Scaling After Visit 2 | 0.83 (0.70) | 0.95 (0.64)
  Patient Diary Pustules After Visit 2 | 0.38 (0.67) | 0.58 (0.75)
  Patient Diary Swelling After Visit 2 | 1.17 (0.90) | 1.04 (0.89)
  Patient Diary Pain After Visit 2 | 0.58 (0.74) | 0.66 (0.74)
  Patient Diary Itch After Visit 2 | 0.56 (0.50) | 1.23 (1.02)
  Patient Diary Burn After Visit 2 | 0.49 (0.66) | 0.65 (0.68)
  Patient Diary Color After Visit 2 | 0.96 (0.81) | 0.64 (0.96)
  Patient Diary Infection After Visit 2 | 0.01 (0.06) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each study visit (spaced 3 months apart) over a period of up to 12 months for each subject.
Description: Systematic assessment is obtained through the principal investigator or sub-investigator asking each subject at each visit for any new illnesses or unexpected events.
Arm/Group | High Energy Treatment Group | Low Energy Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/26
Other Adverse Events (participants affected / at risk) | 7/35 | 7/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Energy Treatment Group (N=35) | Low Energy Placebo Group (N=26)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Concussion (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Basal Cell Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Two raters were used to rate the appearance of the scars. More raters will have been helpful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT02985151/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT02985151/ICF_001.pdf